CLINICAL TRIAL: NCT06274710
Title: Open Access Digital CommunitY Promoting Self-Care, Peer Support, and HEalth LitEracy (ODYSSEE) for Kidney Health (KH) Trial
Brief Title: ODYSSEE Kidney Health Trial
Acronym: ODYSSEE-KH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Scarborough General Hospital (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-5554
Record Dates: First submitted 2023-10-19; First posted 2024-02-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Cognitive behavioural therapy; Motivational interviewing; eHealth; Self-care behaviours; Clinical Trial; Health-related quality of life; Digital health; Digital counselling; Clinical outcomes
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ODYSSEE-KH (Experimental): Participants in the intervention arm of the trial will have full access to digital counselling materials for CKD self-care and RRT education. Program engagement is dynamic with videos, digital handouts, animated charts, infographics, interactive digital trackers, and self-assessment forms. Patients will receive weekly email links to digital sessions (Supplements 1 and 2). Initial sessions will build motivation for therapeutic change. Subsequent sessions follow CBT guidelines. Finally, a monthly video posted on ODYSSEE will address common challenges and patient comments or queries.
  Interventions: Behavioral: ODYSSEE-KH
- Usual care (UC) (No Intervention): UC is the standard of usual care which provides patients with conventional digital CKD education

INTERVENTIONS:
Behavioral: ODYSSEE-KH — Automated digital counselling program
  Arms: ODYSSEE-KH

SUMMARY:
INTRODUCTION

Severe CKD is defined as a risk of greater than 10% for progressing to RRT [home hemodialysis (HHD), home peritoneal dialysis (HPD), and transplantation] within 2 years. There is a need to improve access to CKD self-care counselling and RRT education for patients with severe CKD. Trials of CKD self-care education have achieved therapeutic benefits with moderate to high patient-provider contact. There is high potential for a trial of digital counselling for CKD self-care and RRT education to enhance patient health and quality of life.

HYPOTHESES

The primary hypothesis is that ODYSSEE-KH versus usual care (UC) will significantly increase the incidence of home RRT, measured by a composite index of HHD, HPD, and preemptive kidney transplant at trial completion (median = 19 months; range: 12 to 27 months).

The secondary hypothesis is that ODYSSEE-KH for CKD self-care and RRT education improves Home RRT, RRT preparation, annual hospitalization rate, engagement with CKD self-care resources at months 6 and 12 and trial completion and scores on outcome measures.

RECRUITMENT

Patients diagnosed with CKD who are 18 years of age or older were recruited from University Health Network (UHN), Sunnybrook Hospital, Scarborough Health Network, and The Ottawa Hospital.

DESIGN

ODYSSEE-KH is a double-arm, parallel-group, randomized controlled trial that has assessments at baseline, months 6 and 12, and trial completion (median = 19 months; range: 12 to 27 months). This is a single-blind design with research personnel masked.

ODYSSEE-KH combines automated digital counselling of CKD self-care with renal replacement therapy (RRT) education. UC enhances the standard of usual care by providing patients with conventional digital CKD education. Over 27 months, patients will be emailed on a weekly basis with a digital link to log on to their respective program using a password-protected, personal account.

ANALYSIS

Separate GLMs will evaluate if Digital Counselling versus UC is independently associated with outcomes at months 6 and 12 and trial completion (median = 19; range: 12 to 27 months). Dependent variables include the KDQOL-SF, SF-36, EUROIA, PHQ-9, GAD-7, MIDLS, ESSI, PWB, BMPN, AI, as well as a modified SEMCD-6. Multivariable models will adjust for baseline assessments of each outcome and potential baseline covariates (noted above). In all GLMs, significant interactions will be followed by subgroup analyses with Bonferroni post hoc tests.

DETAILED DESCRIPTION:
BACKGROUND

In Canada, severe CKD prevalence is 14.9 per 1000 persons. The mortality risk is greatest for pre-dialysis patients with stage 4 or 5 CKD (182 deaths per 1000). The annual cost of medical services for Canadians with CKD is $32 billion, with an annual cost per patient of $20 124 and $23 303 at stages 4 and 5, respectively. Persons with stage 4 or 5 CKD also report a lower quality of life and experience the greatest decrement in quality-adjusted life years projected over time.

Kidney transplantation is recognized as the gold standard for RRT due to its benefit for improving clinical outcomes and quality of life. However, the median wait time in Canada for kidney transplantation is 4 years. Approximately 80% of patients with severe CKD are suitable to receive dialysis. Most CKD patients (76%) receive in-center hemodialysis (ICHD), while only 17% receive home hemodialysis (HHD) and 2.5% receive home peritoneal dialysis (HPD). When considering the systemic and patient burden of CKD, it is important to note that ICHD does not offer added survival benefits, and patients who receive home dialysis report greater quality of life. There is also a lower cost for providing HHD and HPD versus ICHD.

Task force statements and reviews advocate for informed patient choice about HHD and HPD, and patients who receive RRT education are more likely to select home dialysis. However, 38% of CKD patients on dialysis report that they were not informed or involved in the decision to select their dialysis modality, and 64% report that education on managing CKD was inadequate or not provided. During the SARS-CoV-2 pandemic, in-hospital dialysis was associated with a 3- to 4-fold increased risk of virus infection and a high mortality rate of 21-34%, which further supports HHD and HPD.

Task force committees concede that patients with severe CKD require specialized nephrology services that include (i) education to promote informed decision-making about RRT and (ii) counselling to improve quality of life and CKD self-care (i.e., attending medical appointments and adhering to medications, dialysis, fluid and dietary guidelines, monitoring symptoms, engaging in an active lifestyle, and refraining from smoking). A Cochrane review of 40 longitudinal cohort studies (pooled N = 63 887) reported that early access to specialized services predicted shorter hospitalization for initial admission [-9.1 days; 95% confidence interval (CI): -11 to -7], and reduced mortality at 12 months (RR =0.65; 95% CI: 0.62 to 0.69) and 5 years (RR = 0.66; 95% CI: 0.60 to 0.71). Corroborating findings from a meta-analysis (pooled N = 648) and a recent randomized trial (N = 130) show that CKD self-care education with telehealth services is associated with reduced hospital admissions and emergency department visits. A further meta-analysis (pooled N = 1647) reported improved quality of life with CKD self-care education or counselling. It is, therefore, vital to commence a CKD self-care and RRT initiative that is evidence-based, scalable, and patient-centred.

RATIONALE

Trials of CKD self-care education have achieved therapeutic benefits with moderate to high patient-provider contact. Direct contact time with individual patients has been estimated in a systematic review of behavioural counselling to range up to 6 hours, which limits the scalability of conventional programs. Moreover, current CKD patient education programs are infrequent and not standardized. CKD patients have reported in several studies that they are not adequately informed or involved in decision-making about their care. In addition, patient barriers that influence informed decision-making about home-based RRT are not adequately addressed. Importantly, patients with severe CKD express marked interest in counselling that extends beyond information about procedures or medical outcomes. Patient interests include ways to improve quality of life and psychosocial well-being, control of care, safety, ability to maintain daily activities, and communication with health care providers. There is high potential for a trial of digital counselling for CKD self-care and RRT education to enhance patient health and quality of life. The risk for mortality decreases in a stepwise manner with incremental adherence to self-care[PR1] . A digital strategy is feasible to promote CKD self-care since 90% of Canadians report internet access, which includes 81 to 93% of persons in the 2 lowest income quartiles, 87% of individuals aged 50 to 64 years, and 66% of those equal to or greater than 65 years.

HYPOTHESES

The primary hypothesis is that ODYSSEE-KH versus UC will significantly increase the incidence of home RRT, measured by a composite index27 of HHD, HPD, and preemptive kidney transplant at trial completion (median = 19 months; range: 12 to 27 months).

The secondary hypothesis is that ODYSSEE-KH versus UC will significantly improve the following:

1. Home RRT (composite index of HHD, HPD, and preemptive kidney transplant at trial completion)27
2. RRT preparation [incidence of arteriovenous fistula (AVF) or arteriovenous graft (AVG), or PD catheter] at trial completion (median = 19 months; range: 12 to 27 months)
3. Annual hospitalization rate, calculated as a rate per patient per year, at trial completion (median = 19 months; range: 12 to 27 months)
4. Engagement with CKD self-care resources at months 6 and 12 and trial completion (median = 19 months; range: 12 to 27 months), defined by the sum of logon minutes, the sum of logons, and the number of logon days prior to a lapse of equal to or greater than 2 months (taken from CHF-CePPORT49-52 and the former pilot study).
5. The following patient-reported outcome measures of HRQL at baseline, months 6 and 12, and trial completion (median = 19 months; range: 12 to 27 months):

   * HRQL (KDQOL-SF and SF-36)
   * Engagement in activities for living well (EUROIA)
   * Depression (PHQ-9)
   * Anxiety (GAD-7)
   * Mattering in life domains (MIDLS)
   * Social support (ESSI)
   * Psychological well-being (PWB)
   * Psychological needs (BMPN)
   * Extrinsic and intrinsic aspirations (AI)
   * Self-efficacy in managing a chronic disease (SEMCD-6)

POTENTIAL RISKS

There is a potential risk that patients in the intervention arm will feel uncomfortable while using ODYSSEE-KH because they are not familiar with the software. Participants may also feel uncomfortable answering certain questions posed in the questionnaire packages, such as those pertaining to mental health, social support, loneliness, and disease burden.

SAFETY PARAMETERS

This is a non-invasive, digital (behavioural) counselling trial. It is complementary in nature and patients will be aware that they can withdraw at any time based on the informed consent procedure. Therefore, there are no significant safety issues associated with this trial.

Personal accounts on the ODYSSEE program will be password-protected. The website itself is hosted on the secure UHN server.

Some of the items presented in the self-report measures of HRQL pertain to mental, physical, social, and occupational functioning. If participants have any concerns about answering one or more questions posed in the questionnaire package, they may contact our office by email or telephone so that their concerns may be addressed. A refusal to respond to any questionnaire item will be accommodated for.

STATISTICAL PLAN

A time-to-event analysis at trial completion (median = 19; range: 12 to 27 months) will be performed using a multivariable Cox Proportional Hazards (PH) model. It will evaluate if Digital Counselling versus UC significantly improves the likelihood for home-based RRT, based on a composite endpoint of first of HPD, HHD, or preemptive kidney transplant. Potential confounders (e.g., age, gender) will be selected using forward (p < 0.05) and backward (p < 0.10) stepwise selection.

A multivariable Cox PH model will assess if Digital Counselling versus UC significantly improves the likelihood for the composite endpoint of incidence of AVF, or AVG, or PD catheter at trial completion (median = 19; range: 12 to 27 months).

At trial completion (median = 19; range: 12 to 27 months), log-linear Poisson models will be conducted for hospitalization rate, per patient, per year. A multivariable Cox PH model will then evaluate if Digital Counselling versus UC significantly increases time to hospitalization.

Separate Generalized Linear Models (GLMs) will evaluate if Digital Counselling versus UC evokes greater CKD self-care program adherence at months 6 and 12- and trial completion (median = 19; range: 12 to 27 months). The dependent variable will be the sum of logon time and the predictors will include age, gender, and trial arm (Digital Counselling or UC), as well as potential baseline confounders (noted above). The GLM for the endpoints will be repeated using the sum of logons as the dependent variable. Finally, for these endpoints, a multivariable Poisson model will evaluate whether Digital Counselling versus UC is associated with greater duration of engagement (defined as the sum of logons, sum of logon hours, and number of logon days prior to a logon lapse of equal to or greater than 1 month), adjusting for sex, age, and potential confounding variables (noted above).

Separate GLMs will evaluate if Digital Counselling versus UC is independently associated with outcomes at months 6 and 12 and trial completion (median = 19; range: 12 to 27 months). Dependent variables include the KDQOL-SF, AI, EUROIA, ESSI, PHQ-9, GAD-7, BMPN, PWB, MIDLS and SF-36, as well as a modified SEMCD-6. Multivariable models will adjust for baseline assessments of each outcome and potential baseline covariates (noted above). In all GLMs, significant interactions will be followed by subgroup analyses with Bonferroni post-hoc tests.

After testing interactions between Digital Counselling versus UC and gender in the primary and secondary outcome analyses, separate exploratory analyses will be performed for gender categories sufficiently represented in the sample. Separate competing risk models will be employed to evaluate time to each of the following outcomes: HPD, HHD, and preemptive kidney transplant.

DEVIATIONS FROM STATISTICAL PLAN

A need to deviate from the original statistical plan is not anticipated because exploratory analyses are included. Nevertheless, the Statistical Analyses and Methodology Committee will be consulted regularly throughout the trial.

SAMPLE SIZE

The sample estimate for the ODYSSEE-KH trial, with monitoring over 19 months, is only 64 patients, type 1 error = 5% and power = 80%.The CKD pilot study achieved moderate program adherence, similar to the CHF-CEPPORT trial whereby the median proportion of sessions access was 61%. The sample estimate to detect this effect with a double-group design, type 1 error of 5%, and power of 80% is N = 114. In sum, the conservative sample estimate used for our primary outcome will ensure appropriate statistical power to evaluate our secondary outcomes of hospitalization and usability. The final sample estimate is N = 344, with a type 1 error of 5% and a power of 80%.

COMPLIANCE

Participation will be supported by senior clinical staff members to ensure that trial activities are presented as complementary to a patient's healthcare. The research team will promote adherence to online assessments via REDCap® with email, telephone, and in-person reminders.

WITHDRAWAL

This trial does not include invasive procedures or changes to medications that could trigger a significant clinical event. Therefore, the need to actively withdraw subjects from this complementary, behavioural (digital) counselling program is not anticipated.

CRITERIA FOR TRIAL TERMINATION

The ODYSSEE-KH trial would have been terminated prematurely in the event of a recurrent adverse event that was related to our trial procedures or content.

QUALITY CONTROL AND ASSURANCE

Daily management and monitoring of recruitment and assessment activities will be completed by the research coordinator.

Responsibility for quality control will remain with the full team. The multidisciplinary research team holds senior administrative, clinical, and research appointments at participating institutions

CONSENT

Initial contact with the patient will be made only by members of the circle of care, who will not attempt to obtain informed consent from the patients. Clinical staff in participating outpatient nephrology clinics will identify patients who meet trial criteria and will obtain verbal consent to be approached by the research team. Informed consent will be obtained either in person or virtually. Regardless of the method, A follow-up email will be sent to the participant by the research team containing the participant's onboarding information (i.e., hyperlink to ODYSSEE platform, username, and temporary password), as well instructions and tutorial videos on how to access the ODYSSEE platform.

In-person, a trained research team member will approach the potential participant during their clinic appointment and will provide them with a hard copy of the Informed Consent Form. The trained research team member will discuss the content of the Informed Consent Form with the patient and will address any questions and/or concerns relating to the trial that the patient may have. Patients will be informed that their participation is voluntary and that it will have no bearing on their healthcare. Moreover, this message is clearly conveyed in the Informed Consent Form. The trained research team member will provide the patient with as much time as they require to make an informed decision about participating in the trial.If the patient decides to consent to participate in the trial, informed consent will be obtained in person via double signatures on hard copies. One copy will be kept on file by the research team and the other copy will be retained by the participant.

Virtually, a trained research team member will contact the patient by telephone to confirm their interest in the trial. The trained research team member will email the patient a hyperlink to the Informed Consent Form, housed on the UHN REDCap server ®. The patient will be asked to refrain from signing the Informed Consent Form until they have had an opportunity to discuss the trial, as well as any questions and/or concerns they may have, with the research team. The trained research team member will discuss the content of the Informed Consent Form with the patient over the telephone and will address any questions and/or concerns relating to the trial that the patient may have. Patients will be informed that their participation is voluntary and that it will have no bearing on their healthcare. Moreover, this message is clearly conveyed in the Informed Consent Form. The trained research team member will provide the patient with as much time as they require to make an informed decision about participating in the trial. If the patient decides to consent to participate in the trial, informed consent will be obtained virtually via electronic signatures on PDF copies. A copy will be kept on file by the research team and the other copy will be sent to the participant by email.

DATA STORAGE

All data will be stored on secure servers within the UHN digital environment, ensuring that security measures are well-developed to protect the data from external intrusion. Data will be stored for 10 years as per UHN Research procedure.

The digital forms and materials will be retained on the secure UHN server for at least 10 years from the completion of the trial.

Data will be available from the corresponding author pending approval of research ethics boards of participating institutions and on a reasonable request received from qualified researchers trained in human subject confidentiality protocols.

PRIVACY AND CONFIDENTIALITY

Subjects are issued a tracking number when data involving identifying information is transmitted for analysis. Subject anonymity and confidentiality have been preserved. Only aggregate data will be published.

All research personnel have signed an employee confidentiality agreement ensuring that confidential information is not disclosed to any other person or entity. All source documents containing personal identifiers are stored in filing cabinets under lock and key. The database is stored electronically on the firewall-protected server, making it inaccessible externally. Access to the room containing the research file server is restricted to designated persons who are employed by the Behavioural Cardiology Research Unit at the UHN.

Discussion of the trial with persons outside the research team will never reveal the personal identifiers of participants. All-access to data is denied to persons outside the research team. Data transmission occurs via encrypted storage material over the Internet.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients who are at least 18 years old, that have a greater than a 10% risk of requiring dialysis within 2 years, using the 4-variable 2-year Kidney Failure Risk Equation,1,2 and are registered in a nephrology clinic (including an in-center dialysis clinic) at a participating hospital
* Confirmation from a referring nephrologist that the CKD has been stable for at least 1 month at the time of enrollment
* Oral and written comprehension of English or French
* Informed written consent
* At least a basic level of self-reported computer literacy
* Access to the internet and a computer

Exclusion Criteria:

* Previous kidney transplant or waitlisted for organ transplant at the time of enrollment
* Severe co-morbidities that prohibit full participation (e.g., dementia, clinically severe depression)
* Diagnosis of a medical condition for which the life expectancy is less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of home RRT | Trial completion (median = 19 months, range = 12-27 months)
  The primary objective is to determine whether an automated digital counselling program for CKD self-care and RRT education improves RRT or preemptive renal transplant over a median of 19 months. As in our previous research,45-47 assessment of RRT includes documentation of incident home dialysis (HPD or HHD) or preemptive kidney transplant (before dialysis) in a composite index, using data from the Canadian Institute for Health Information (CIHI).48

SECONDARY OUTCOMES:
Improvement of Home RRT | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  The secondary objective is to determine whether an automated digital counselling program for CKD self-care and RRT education improves home RRT (measured by a composite index of documented HHD, HPD, or pre-emptive kidney transplantation)
Improvement of RRT preparation with planned dialysis access | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  RRT preparation with planned dialysis access, based on the incidence of arteriovenous fistula (AVF), arteriovenous graft (AVG), or peritoneal dialysis (PD) catheter
Incidence of annual hospitalization rate | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Obtained using CIHI databases,48 assessed as the rate, per patient, per year, and defined from date of randomization to the earliest of death, start of dialysis
Engagement with RRT education and CKD self-care counselling resources | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Measured by the sum of logons, sum of logon hours, and number of logon days prior to a logon lapse of equal to or greater than 1 month (data is obtained using backend analytic tools of ODYSSEE, as in CHF-CePPORT49-52 and the previous pilot study)53-55
Self-reported engagement in activities for living well | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Evaluation of Goal-Directed Activities to Promote Well-Being and Health (EUROIA), developed by the principal investigator
Self-reported assessment for health-related quality of life due to kidney disease | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  36-Item Kidney Disease Quality of Life - Short Form (KDQOL-SF)
Self-reported assessment of people's aspirations and goals | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Aspirations Index (AI)
Self-reported measure of overall health (e.g. pain, mental health, physical, role and social functioning) | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  36-Item Short Form (SF-36)
Self-reported depression | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  9-Item Patient Health Questionnaire (PHQ-9)
Self-reported perceived social support | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  ENRICHD Social Support Instrument (ESSI)
Self-reported psychological wellbeing | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Flourishing Scale (FS)
Self-reported anxiety | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  7-Item Generalized Anxiety Disorder instrument (GAD-7)
Self-reported feeling of value to self and others | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  9-Item Mattering in Domains of Life Scale (MIDLS)
Self-reported measure of psychological wellbeing and happiness | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  18-Item Psychological Wellbeing Scale (PWB)
Self-reported measure of overall life experience | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  18-Item Balanced Measure of Psychological Needs (BMPN)
Self-reported measure of well-being | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  WHO-5 Item Well-Being Index
Self-reported readiness for change (motivation) | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Patient-reported readiness to initiate renal replacement therapy
Self-reported confidence in doing life activities | Month 6, month 12, Trial completion (median = 19 months, range = 12-27 months)
  Self-Efficacy for Managing Chronic Diseases 6-item Scale (SEMCD-6)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nolan, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tangri N, Stevens LA, Griffith J, Tighiouart H, Djurdjev O, Naimark D, Levin A, Levey AS. A predictive model for progression of chronic kidney disease to kidney failure. JAMA. 2011 Apr 20;305(15):1553-9. doi: 10.1001/jama.2011.451. Epub 2011 Apr 11. PMID 21482743
- [Background] Tangri N, Grams ME, Levey AS, Coresh J, Appel LJ, Astor BC, Chodick G, Collins AJ, Djurdjev O, Elley CR, Evans M, Garg AX, Hallan SI, Inker LA, Ito S, Jee SH, Kovesdy CP, Kronenberg F, Heerspink HJ, Marks A, Nadkarni GN, Navaneethan SD, Nelson RG, Titze S, Sarnak MJ, Stengel B, Woodward M, Iseki K; CKD Prognosis Consortium. Multinational Assessment of Accuracy of Equations for Predicting Risk of Kidney Failure: A Meta-analysis. JAMA. 2016 Jan 12;315(2):164-74. doi: 10.1001/jama.2015.18202. PMID 26757465
- [Background] Bello AK, Ronksley PE, Tangri N, Kurzawa J, Osman MA, Singer A, Grill A, Nitsch D, Queenan JA, Wick J, Lindeman C, Soos B, Tuot DS, Shojai S, Brimble S, Mangin D, Drummond N. Prevalence and Demographics of CKD in Canadian Primary Care Practices: A Cross-sectional Study. Kidney Int Rep. 2019 Jan 21;4(4):561-570. doi: 10.1016/j.ekir.2019.01.005. eCollection 2019 Apr. PMID 30993231
- [Background] Manns B, Hemmelgarn B, Tonelli M, Au F, So H, Weaver R, Quinn AE, Klarenbach S; for Canadians Seeking Solutions and Innovations to Overcome Chronic Kidney Disease. The Cost of Care for People With Chronic Kidney Disease. Can J Kidney Health Dis. 2019 Apr 4;6:2054358119835521. doi: 10.1177/2054358119835521. eCollection 2019. PMID 31057803
- [Background] Inker LA, Astor BC, Fox CH, Isakova T, Lash JP, Peralta CA, Kurella Tamura M, Feldman HI. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for the evaluation and management of CKD. Am J Kidney Dis. 2014 May;63(5):713-35. doi: 10.1053/j.ajkd.2014.01.416. Epub 2014 Mar 16. PMID 24647050
- [Background] Gorodetskaya I, Zenios S, McCulloch CE, Bostrom A, Hsu CY, Bindman AB, Go AS, Chertow GM. Health-related quality of life and estimates of utility in chronic kidney disease. Kidney Int. 2005 Dec;68(6):2801-8. doi: 10.1111/j.1523-1755.2005.00752.x. PMID 16316356
- [Background] Landreneau K, Lee K, Landreneau MD. Quality of life in patients undergoing hemodialysis and renal transplantation--a meta-analytic review. Nephrol Nurs J. 2010 Jan-Feb;37(1):37-44. PMID 20333902
- [Background] Vinson AJ, Perl J, Tennankore KK. Survival Comparisons of Home Dialysis Versus In-Center Hemodialysis: A Narrative Review. Can J Kidney Health Dis. 2019 Jul 13;6:2054358119861941. doi: 10.1177/2054358119861941. eCollection 2019. PMID 31321065
- [Background] Eneanya ND, Maddux DW, Reviriego-Mendoza MM, Larkin JW, Usvyat LA, van der Sande FM, Kooman JP, Maddux FW. Longitudinal patterns of health-related quality of life and dialysis modality: a national cohort study. BMC Nephrol. 2019 Jan 8;20(1):7. doi: 10.1186/s12882-018-1198-5. PMID 30621634
- [Background] Klarenbach S, Tonelli M, Pauly R, Walsh M, Culleton B, So H, Hemmelgarn B, Manns B. Economic evaluation of frequent home nocturnal hemodialysis based on a randomized controlled trial. J Am Soc Nephrol. 2014 Mar;25(3):587-94. doi: 10.1681/ASN.2013040360. Epub 2013 Nov 14. PMID 24231665
- [Background] Chan CT, Wallace E, Golper TA, Rosner MH, Seshasai RK, Glickman JD, Schreiber M, Gee P, Rocco MV. Exploring Barriers and Potential Solutions in Home Dialysis: An NKF-KDOQI Conference Outcomes Report. Am J Kidney Dis. 2019 Mar;73(3):363-371. doi: 10.1053/j.ajkd.2018.09.015. Epub 2018 Dec 10. PMID 30545707
- [Background] Dahlerus C, Quinn M, Messersmith E, Lachance L, Subramanian L, Perry E, Cole J, Zhao J, Lee C, McCall M, Paulson L, Tentori F. Patient Perspectives on the Choice of Dialysis Modality: Results From the Empowering Patients on Choices for Renal Replacement Therapy (EPOCH-RRT) Study. Am J Kidney Dis. 2016 Dec;68(6):901-910. doi: 10.1053/j.ajkd.2016.05.010. Epub 2016 Jun 21. PMID 27337991
- [Background] Akbari A, Clase CM, Acott P, Battistella M, Bello A, Feltmate P, Grill A, Karsanji M, Komenda P, Madore F, Manns BJ, Mahdavi S, Mustafa RA, Smyth A, Welcher ES. Canadian Society of Nephrology commentary on the KDIGO clinical practice guideline for CKD evaluation and management. Am J Kidney Dis. 2015 Feb;65(2):177-205. doi: 10.1053/j.ajkd.2014.10.013. Epub 2014 Nov 4. PMID 25511161
- [Background] Smart NA, Dieberg G, Ladhani M, Titus T. Early referral to specialist nephrology services for preventing the progression to end-stage kidney disease. Cochrane Database Syst Rev. 2014 Jun 18;(6):CD007333. doi: 10.1002/14651858.CD007333.pub2. PMID 24938824
- [Background] He T, Liu X, Li Y, Wu Q, Liu M, Yuan H. Remote home management for chronic kidney disease: A systematic review. J Telemed Telecare. 2017 Jan;23(1):3-13. doi: 10.1177/1357633X15626855. Epub 2016 Jul 9. PMID 27269795
- [Background] Fishbane S, Agoritsas S, Bellucci A, Halinski C, Shah HH, Sakhiya V, Balsam L. Augmented Nurse Care Management in CKD Stages 4 to 5: A Randomized Trial. Am J Kidney Dis. 2017 Oct;70(4):498-505. doi: 10.1053/j.ajkd.2017.02.366. Epub 2017 Apr 7. PMID 28396108
- [Background] Lin MY, Liu MF, Hsu LF, Tsai PS. Effects of self-management on chronic kidney disease: A meta-analysis. Int J Nurs Stud. 2017 Sep;74:128-137. doi: 10.1016/j.ijnurstu.2017.06.008. Epub 2017 Jun 21. PMID 28689160
- [Background] Fadem SZ, Walker DR, Abbott G, Friedman AL, Goldman R, Sexton S, Buettner K, Robinson K, Peters TG. Satisfaction with renal replacement therapy and education: the American Association of Kidney Patients survey. Clin J Am Soc Nephrol. 2011 Mar;6(3):605-12. doi: 10.2215/CJN.06970810. Epub 2011 Feb 17. PMID 21330485
- [Background] Walker RC, Hanson CS, Palmer SC, Howard K, Morton RL, Marshall MR, Tong A. Patient and caregiver perspectives on home hemodialysis: a systematic review. Am J Kidney Dis. 2015 Mar;65(3):451-63. doi: 10.1053/j.ajkd.2014.10.020. Epub 2015 Jan 10. PMID 25582285
- [Background] Khaw KT, Wareham N, Bingham S, Welch A, Luben R, Day N. Combined impact of health behaviours and mortality in men and women: the EPIC-Norfolk prospective population study. PLoS Med. 2008 Jan 8;5(1):e12. doi: 10.1371/journal.pmed.0050012. PMID 18184033
- [Background] Simpson SH, Eurich DT, Majumdar SR, Padwal RS, Tsuyuki RT, Varney J, Johnson JA. A meta-analysis of the association between adherence to drug therapy and mortality. BMJ. 2006 Jul 1;333(7557):15. doi: 10.1136/bmj.38875.675486.55. Epub 2006 Jun 21. PMID 16790458
- [Background] Kummervold PE, Chronaki CE, Lausen B, Prokosch HU, Rasmussen J, Santana S, Staniszewski A, Wangberg SC. eHealth trends in Europe 2005-2007: a population-based survey. J Med Internet Res. 2008 Nov 17;10(4):e42. doi: 10.2196/jmir.1023. PMID 19017584
- [Background] Milazi M, Bonner A, Douglas C. Effectiveness of educational or behavioral interventions on adherence to phosphate control in adults receiving hemodialysis: a systematic review. JBI Database System Rev Implement Rep. 2017 Apr;15(4):971-1010. doi: 10.11124/JBISRIR-2017-003360. PMID 28398983
- [Background] Hung CS, Lee J, Chen YH, Huang CC, Wu VC, Wu HW, Chuang PY, Ho YL. Effect of Contract Compliance Rate to a Fourth-Generation Telehealth Program on the Risk of Hospitalization in Patients With Chronic Kidney Disease: Retrospective Cohort Study. J Med Internet Res. 2018 Jan 24;20(1):e23. doi: 10.2196/jmir.8914. PMID 29367185
- [Background] Beishuizen CR, Stephan BC, van Gool WA, Brayne C, Peters RJ, Andrieu S, Kivipelto M, Soininen H, Busschers WB, Moll van Charante EP, Richard E. Web-Based Interventions Targeting Cardiovascular Risk Factors in Middle-Aged and Older People: A Systematic Review and Meta-Analysis. J Med Internet Res. 2016 Mar 11;18(3):e55. doi: 10.2196/jmir.5218. PMID 26968879
- [Background] Garcia-Lizana F, Sarria-Santamera A. New technologies for chronic disease management and control: a systematic review. J Telemed Telecare. 2007;13(2):62-8. doi: 10.1258/135763307780096140. PMID 17359568
- [Background] Comellas M, Walker EA, Movsas S, Merkin S, Zonszein J, Strelnick H. Training community health promoters to implement diabetes self-management support programs for urban minority adults. Diabetes Educ. 2010 Jan-Feb;36(1):141-51. doi: 10.1177/0145721709354606. Epub 2009 Dec 4. PMID 19966071
- [Background] Clark AM, Hartling L, Vandermeer B, McAlister FA. Meta-analysis: secondary prevention programs for patients with coronary artery disease. Ann Intern Med. 2005 Nov 1;143(9):659-72. doi: 10.7326/0003-4819-143-9-200511010-00010. PMID 16263889
- [Background] Hunting G, Shahid N, Sahakyan Y, Fan I, Moneypenny CR, Stanimirovic A, North T, Petrosyan Y, Krahn MD, Rac VE. A multi-level qualitative analysis of Telehomecare in Ontario: challenges and opportunities. BMC Health Serv Res. 2015 Dec 9;15:544. doi: 10.1186/s12913-015-1196-2. PMID 26645639
- [Background] Pechlivanoglou P, Abrahamyan L, MacKeigan L, Consiglio GP, Dolovich L, Li P, Cadarette SM, Rac VE, Shin J, Krahn M. Factors affecting the delivery of community pharmacist-led medication reviews: evidence from the MedsCheck annual service in Ontario. BMC Health Serv Res. 2016 Nov 21;16(1):666. doi: 10.1186/s12913-016-1888-2. PMID 27871324
- [Background] Slater M, Bielecki J, Alba AC, Abrahamyan L, Tomlinson G, Mak S, MacIver J, Zieroth S, Lee D, Wong W, Krahn M, Ross H, Rac VE. Comparative effectiveness of the different components of care provided in heart failure clinics-protocol for a systematic review and network meta-analysis. Syst Rev. 2019 Feb 2;8(1):40. doi: 10.1186/s13643-019-0953-4. PMID 30711016
- [Background] Nolan RP, Payne AY, Ross H, White M, D'Antono B, Chan S, Barr SI, Gwadry-Sridhar F, Nigam A, Perreault S, Farkouh M, McDonald M, Goodman J, Thomas S, Zieroth S, Isaac D, Oh P, Rajda M, Chen M, Eysenbach G, Liu S, Zbib A. An Internet-Based Counseling Intervention With Email Reminders that Promotes Self-Care in Adults With Chronic Heart Failure: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2014 Jan 30;3(1):e5. doi: 10.2196/resprot.2957. PMID 24480783
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Mitchell PH, Powell L, Blumenthal J, Norten J, Ironson G, Pitula CR, Froelicher ES, Czajkowski S, Youngblood M, Huber M, Berkman LF. A short social support measure for patients recovering from myocardial infarction: the ENRICHD Social Support Inventory. J Cardiopulm Rehabil. 2003 Nov-Dec;23(6):398-403. doi: 10.1097/00008483-200311000-00001. No abstract available. PMID 14646785
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Ryff CD. In the eye of the beholder: views of psychological well-being among middle-aged and older adults. Psychol Aging. 1989 Jun;4(2):195-201. doi: 10.1037//0882-7974.4.2.195. PMID 2789747
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Nolan RP, Feldman R, Dawes M, Kaczorowski J, Lynn H, Barr SI, MacPhail C, Thomas S, Goodman J, Eysenbach G, Liu S, Tanaka R, Surikova J. Randomized Controlled Trial of E-Counseling for Hypertension: REACH. Circ Cardiovasc Qual Outcomes. 2018 Jul;11(7):e004420. doi: 10.1161/CIRCOUTCOMES.117.004420. PMID 30006474
- [Background] Nolan RP, Liu S, Feldman R, Dawes M, Barr S, Lynn H, Gwardy-Sridhar F, Thomas SG, Goodman J, Oh P, Kaczorowski J, Chessex C, Hachinski V, Shoemaker K. Reducing risk with e-based support for adherence to lifestyle change in hypertension (REACH): protocol for a multicentred randomised controlled trial. BMJ Open. 2013 Aug 21;3(8):e003547. doi: 10.1136/bmjopen-2013-003547. PMID 23965936
- [Background] Liu S, Tanaka R, Barr S, Nolan RP. Effects of self-guided e-counseling on health behaviors and blood pressure: Results of a randomized trial. Patient Educ Couns. 2020 Mar;103(3):635-641. doi: 10.1016/j.pec.2019.10.007. Epub 2019 Oct 19. PMID 31669047
- [Background] United States Renal Data System. 2022 USRDS Annual Data Report: Epidemiology of kidney disease in the United States. (National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD).
- [Background] Nguyen NTQ, Cockwell P, Maxwell AP, Griffin M, O'Brien T, O'Neill C. Chronic kidney disease, health-related quality of life and their associated economic burden among a nationally representative sample of community dwelling adults in England. PLoS One. 2018 Nov 26;13(11):e0207960. doi: 10.1371/journal.pone.0207960. eCollection 2018. PMID 30475893
- [Background] Information, C. I. f. H. Annual statistics on organ replacement in Canada, 2011 to 2020. (2021).
- [Background] Mendelssohn DC, Mujais SK, Soroka SD, Brouillette J, Takano T, Barre PE, Mittal BV, Singh A, Firanek C, Story K, Finkelstein FO. A prospective evaluation of renal replacement therapy modality eligibility. Nephrol Dial Transplant. 2009 Feb;24(2):555-61. doi: 10.1093/ndt/gfn484. Epub 2008 Aug 28. PMID 18755848
- [Background] Krahn MD, Bremner KE, de Oliveira C, Dixon SN, McFarlane P, Garg AX, Mitsakakis N, Blake PG, Harvey R, Pechlivanoglou P. Home Dialysis Is Associated with Lower Costs and Better Survival than Other Modalities: A Population-Based Study in Ontario, Canada. Perit Dial Int. 2019 Nov-Dec;39(6):553-561. doi: 10.3747/pdi.2018.00268. Epub 2019 Oct 3. PMID 31582466
- [Background] Trinh E, Chan CT, Perl J. Dialysis modality and survival: Done to death. Semin Dial. 2018 Jul;31(4):315-324. doi: 10.1111/sdi.12692. Epub 2018 Mar 14. PMID 29539161
- [Background] Ludlow MJ, George CR, Hawley CM, Mathew TH, Agar JW, Kerr PG, Lauder LA. How Australian nephrologists view home dialysis: results of a national survey. Nephrology (Carlton). 2011 May;16(4):446-52. doi: 10.1111/j.1440-1797.2010.01403.x. PMID 21518119
- [Background] Kutner NG, Zhang R, Huang Y, Wasse H. Patient awareness and initiation of peritoneal dialysis. Arch Intern Med. 2011 Jan 24;171(2):119-24. doi: 10.1001/archinternmed.2010.361. Epub 2010 Sep 27. PMID 20876396
- [Background] Van Biesen W, van der Veer SN, Murphey M, Loblova O, Davies S. Patients' perceptions of information and education for renal replacement therapy: an independent survey by the European Kidney Patients' Federation on information and support on renal replacement therapy. PLoS One. 2014 Jul 31;9(7):e103914. doi: 10.1371/journal.pone.0103914. eCollection 2014. PMID 25079071
- [Background] Brunori G, Reboldi G, Aucella F. Lessons Learnt during the COVID-19 Pandemic: For Patients with End-Stage Renal Disease, We Should Prioritize Home-Based Treatment and Telemedicine. Kidney Blood Press Res. 2021;46(1):11-16. doi: 10.1159/000512629. Epub 2021 Jan 29. PMID 33517338
- [Background] Andrassy KM. Comments on 'KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease'. Kidney Int. 2013 Sep;84(3):622-3. doi: 10.1038/ki.2013.243. No abstract available. PMID 23989362
- [Background] Walker AMN, Drozd M, Hall M, Patel PA, Paton M, Lowry J, Gierula J, Byrom R, Kearney L, Sapsford RJ, Witte KK, Kearney MT, Cubbon RM. Prevalence and Predictors of Sepsis Death in Patients With Chronic Heart Failure and Reduced Left Ventricular Ejection Fraction. J Am Heart Assoc. 2018 Oct 16;7(20):e009684. doi: 10.1161/JAHA.118.009684. PMID 30371261
- [Background] Granger BB, Swedberg K, Ekman I, Granger CB, Olofsson B, McMurray JJ, Yusuf S, Michelson EL, Pfeffer MA; CHARM investigators. Adherence to candesartan and placebo and outcomes in chronic heart failure in the CHARM programme: double-blind, randomised, controlled clinical trial. Lancet. 2005 Dec 10;366(9502):2005-11. doi: 10.1016/S0140-6736(05)67760-4. PMID 16338449
- [Background] Bramley TJ, Gerbino PP, Nightengale BS, Frech-Tamas F. Relationship of blood pressure control to adherence with antihypertensive monotherapy in 13 managed care organizations. J Manag Care Pharm. 2006 Apr;12(3):239-45. doi: 10.18553/jmcp.2006.12.3.239. PMID 16623608
- [Background] Authority, C. I. R. Canada's Internet Factbook 2018: Canada's source for current internet data. (2018).
- [Background] Center, P. R. Internet/Broadband Fact Sheet, <https://www.pewresearch.org/internet/fact-sheet/internet-broadband/> (2021).
- [Background] (CIHI), C. I. f. H. I. CIHI, <https://www.cihi.ca/en>
- [Background] Nolan RP, Ross HJ, Farkouh ME, Huszti E, Chan S, Toma M, D'Antono B, White M, Thomas S, Barr SI, Perreault S, McDonald M, Zieroth S, Isaac D, Wielgosz A, Mielniczuk LM. Automated E-Counseling for Chronic Heart Failure: CHF-CePPORT Trial. Circ Heart Fail. 2021 Jan;14(1):e007073. doi: 10.1161/CIRCHEARTFAILURE.120.007073. Epub 2021 Jan 19. PMID 33464959
- [Background] Fezza, G., Sansone, S., Surikova, J., Ross, H. & Nolan, R. Patient Engagement with an Ecounseling Platform is Enhanced Over 12 Months in the CHF-CePPORT Trial. Canadian Journal of Cardiology 34, S148-S149 (2018). https://doi.org:10.1016/j.cjca.2018.07.184
- [Background] Payne AY, Surikova J, Liu S, Ross H, Mechetiuc T, Nolan RP. Usability Testing of an Internet-Based e-Counseling Platform for Adults With Chronic Heart Failure. JMIR Hum Factors. 2015 May 8;2(1):e7. doi: 10.2196/humanfactors.4125. PMID 27026267
- [Background] Wong JV, Yang GJ, Auguste BL, Ong SW, Logan AG, Chan CT, Nolan RP. Automated Digital Counseling Program (ODYSSEE-Kidney Health): A Pilot Study on Health-Related Quality of Life. Kidney360. 2023 Oct 1;4(10):1397-1406. doi: 10.34067/KID.0000000000000229. Epub 2023 Aug 14. PMID 37578528
- [Background] Hays, R. D. et al. Kidney disease quality of life short form (KDQOL-SF™), version 1.3: a manual for use and scoring. Santa Monica, CA: Rand 7994 (1997).
- [Background] Kasser, T., & Ryan, R. M. Aspiration Index [Database record]. APA PsycTests (1993).
- [Background] Sheldon, K. M. & Hilpert, J. C. The balanced measure of psychological needs (BMPN) scale: An alternative domain general measure of need satisfaction. Motivation and Emotion 36, 439-451 (2012). https://doi.org:10.1007/s11031-012-9279-4
- [Background] Scarpa MP, Zopluoglu C, Prilleltensky I. Assessing multidimensional mattering: Development and exploratory validation of the Mattering in Domains of Life Scale (MIDLS). J Community Psychol. 2022 Apr;50(3):1430-1453. doi: 10.1002/jcop.22725. Epub 2021 Oct 4. PMID 34561863
- [Background] (CIHI), C. I. f. H. I. What is the data request process at CIHI?, <https://www.cihi.ca/en/faq/what-is-the-data-request-process-at-cihi>
- [Background] Network, O. R. Living with Chronic Kidney Disease, <https://www.ontariorenalnetwork.ca/en/kidney-care-resources/living-with-chronic-kidney-disease>
- [Background] Foundation, K. Living with Kidney Failure, <https://kidney.ca/Kidney-Health/Living-With-Kidney-Failure> (
- [Background] Miller, W. R. & Rollnick, S. Motivational interviewing: Helping people change, 3rd edition. (Guilford Press, 2013).
- [Background] Weddington, W. W., Jr. Facilitating Treatment Adherence: A Practitioner's Guidebook. JAMA 260, 273-273 (1988). https://doi.org:10.1001/jama.1988.03410020139051
- [Background] (CIHI), C. I. f. H. I. About CIHI, <https://www.cihi.ca/en/about-cihi> (
- [Background] Trinh E, Hanley JA, Nadeau-Fredette AC, Perl J, Chan CT. A comparison of technique survival in Canadian peritoneal dialysis and home hemodialysis patients. Nephrol Dial Transplant. 2019 Nov 1;34(11):1941-1949. doi: 10.1093/ndt/gfz075. PMID 31329952